CLINICAL TRIAL: NCT06514014
Title: Transition From Donor Milk: a Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Brian Stansfield, Professor and Vice Chair for Research, Augusta University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2193903
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-04

CONDITIONS: Preterm Birth; Nutrition, Healthy
Keywords: newborn; human milk
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Open Label Randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor Milk (No Intervention)
- Preterm Infant Formula (Active Comparator)
  Interventions: Dietary Supplement: Preterm Infant Formula

INTERVENTIONS:
Dietary Supplement: Preterm Infant Formula — Transition from donor human milk to preterm infant formula
  Arms: Preterm Infant Formula

SUMMARY:
Preterm and very low birth weight (VLBW, < 1,500g) infants who receive donor human milk (DHM) often experience slow postnatal growth and no clinical data is available to guide the duration of DHM for preterm infants. The investigators hypothesize that transitioning from DHM to preterm infant formula after the first month of life is both safe and conveys improved weight and length gains and fat free mass accumulation.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 1,250 grams
2. At least 28 days of life
3. Diet consisting of donor human milk with/without mother's own milk

Exclusion Criteria:

1. Birth weight below the 5th percentile
2. History of necrotizing enterocolitis, spontaneous intestinal perforation, or other gastrointestinal disorder
3. Congenital anomalies
4. Care team discretion

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight Velocity | 36 weeks post menstrual age
  Weight velocity between birth and 36 weeks post menstrual age
Fat free mass | 36 weeks post menstrual age
  Fat free mass at 36 weeks post menstrual age

SECONDARY OUTCOMES:
Number of Patients with Bronchopulmonary dysplasia | 36 weeks post menstrual age
Number of Patients with Retinopathy of prematurity | 36 weeks post menstrual age
Number of Patients with Sepsis | 36 weeks post menstrual age
Number of Patients with Necrotizing enterocolitis | 36 weeks post menstrual age

CONTACTS AND LOCATIONS:
Locations (1):
- Wellstar-MCG, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No